CLINICAL TRIAL: NCT06582602
Title: A Single Dose Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of Intravenous Infusion and Intravenous Bolus Administration of MK-2060 in Healthy Participants
Brief Title: A Study of MK-2060 in Healthy Participants (MK-2060-016)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 2060-016; MK-2060-016 (Other: MSD)
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Panel A: MK-2060 IV (20 minutes) (Experimental): Participants will receive a single dose of MK-2060 via intravenous (IV) infusion over 20 minutes on Day 1.
  Interventions: Biological: MK-2060
- Panel B: MK-2060 IV (10 minutes) (Experimental): Participants will receive a single dose of MK-2060 via IV infusion over 10 minutes on Day 1.
  Interventions: Biological: MK-2060
- Panel C: MK-2060 IV (5 minutes) (Experimental): Participants will receive a single dose of MK-2060 via syringe over 5 minutes on Day 1.
  Interventions: Biological: MK-2060
- Panel D: MK-2060 IV (2.5 minutes) (Experimental): Participants will receive a single dose of MK-2060 via syringe over 2.5 minutes on Day 1.
  Interventions: Biological: MK-2060
- Panel E: MK-2060 IV (1 minute) (Experimental): Participants will receive a single dose of MK-2060 via syringe over 1 minute on Day 1.
  Interventions: Biological: MK-2060
- Placebo (Placebo Comparator): Participants will receive a single dose of saline via IV infusion or syringe over MK-2060-matched time period on Day 1.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MK-2060 — Single doses of MK-2060 will be administered via IV infusion or syringe on Day 1 according to randomization.
  Arms: Panel A: MK-2060 IV (20 minutes); Panel B: MK-2060 IV (10 minutes); Panel C: MK-2060 IV (5 minutes); Panel D: MK-2060 IV (2.5 minutes); Panel E: MK-2060 IV (1 minute)
Biological: Placebo — Single doses of placebo will be administered via IV infusion or syringe on Day 1 according to randomization.
  Arms: Placebo

SUMMARY:
The goal of the study is to learn about the safety of MK-2060 and if people tolerate it when MK-2060 is given in different forms.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health before randomization
* Has a body mass index (BMI) between ≥18 and ≤32 kg/m^2, inclusive

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has a history of cancer

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants With An Adverse Event (AE) | Up to 134 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants that experience an AE will be reported.
Number of Participants Discontinuing the Study Due to an AE | Up to 134 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants that discontinue the study due to an AE will be reported.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve of MK-2060 From Time 0 to Infinity (AUC0-inf) | Predose and at designated time points post dose up to 120 days
  Plasma samples will be collected at pre-specified time points pre- and post-dose to assess AUC0-inf.
Maximum Observed Plasma Concentration (Cmax) of MK-2060 | Predose and at designated time points post dose up to 120 days
  Plasma samples will be collected at pre-specified time points pre- and post-dose to assess Cmax.
Area Under the Plasma Concentration-Time Curve of MK-2060 From Time 0 to 168 Hours (AUC0-168) | Predose and at designated time points post dose up to 120 days
  Plasma samples will be collected at pre-specified time points pre- and post-dose to assess AUC0-168 hours.
Plasma Concentration of MK-2060 at 168 Hours (C168) | Predose and at designated time points post dose up to 120 days
  Plasma samples will be collected at pre-specified time points pre- and post-dose to assess C168 hours.
Time to Maximum Observed Plasma Drug Concentration (Tmax) of MK-2060 | Predose and at designated time points post dose up to 120 days
  Plasma samples will be collected at pre-specified time points pre- and post-dose to assess Tmax.
Plasma Elimination Terminal Half-life (t ½) of MK-2060 | Predose and at designated time points post dose up to 120 days
  Plasma samples will be collected at pre-specified time points pre- and post-dose to assess t½ .
Apparent Oral Clearance (CL/F) of MK-2060 | Predose and at designated time points post dose up to 120 days
  Plasma samples will be collected at pre-specified time points pre- and post-dose to assess CL/F.
Plasma Apparent Volume of Distribution (Vz/F) of MK-2060 | Predose and at designated time points post dose up to 120 days
  Plasma samples will be collected at pre-specified time points pre- and post-dose to assess Vz/F.
Fold Change From Baseline in Activated Partial Thromboplastin Time (aPTT) of MK-2060 | Baseline and up to 120 days
  Plasma samples will be collected at baseline and pre-specified time points post-dose to assess aPTT values. The fold change from baseline will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Advanced Pharma CR, LLC ( Site 0002), Miami, Florida
  - Alliance for Multispecialty Research, LLC ( Site 0001), Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com